CLINICAL TRIAL: NCT00360594
Title: Initiating Acamprosate Within Versus Post-detoxification in the Rehabilitative Treatment of Alcohol Dependence.
Brief Title: Acamprosate Initiated During Alcohol Detoxification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Helen Pettinati, Ph.D., University of Pennsylvania Treatment Research Cener
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804481; P50DA012756-07 (NIH); CMP-MD-08; DPMC (Other: NIDA)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2010-06

CONDITIONS: Alcohol Use Disorder
Keywords: alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Acamprosate
  Interventions: Drug: Acamprosate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acamprosate — 3 pills (666 mg) for 1998mg/day
  Other Names: Campral
  Arms: 1
Drug: Placebo — 3 pills (666mg) for 1998mg/day
  Arms: 2

SUMMARY:
Acamprosate is approved by the Food and Drug Administration (FDA) for the treatment of alcoholism. The purpose of this study is to see if initiating acamprosate early in alcohol detoxification instead of waiting until detoxification has been completed effects the course of detoxification, adverse events during detoxification, drop out rate during the rehabilitative treatment phase, or overall efficacy of acamprosate for those with alcohol dependence who plan to receive at least two months of rehabilitative pharmacotherapy with acamprosate.

DETAILED DESCRIPTION:
Biphasic clinical trial, consisting of a randomized, double-blind, placebo-controlled detoxification treatment phase (DP), followed by 9-week open-label rehabilitative treatment phase (RP).

ELIGIBILITY:
Inclusion Criteria for Detoxification Treatment Phase

1. Males and females from the ages of 18 to 70 years old. Subjects over the age of 70 years old will be included at the discretion of the PI, with the expectation that these subjects should comprise of no more than 5% of the subjects.
2. Diagnosis of current alcohol dependence according to DSM-IV criteria [DSM-IV criteria will be determined by utilizing the Mini International Neuropsychiatric Interview (MINI)].
3. If necessary, can be medically detoxified in the outpatient setting, as determined by a medical clinician.
4. Meets the following drinking criteria, measured by TLFB: a. reports a minimum of 48 standard alcoholic drinks (avg 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting pharmacotherapy, b. has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males and 4 or more drinks per day in females) within 30 days of starting pharmacotherapy treatment and c. has had a drink within 48 hours of the intake/screening visit or has a CIWA score equal to or greater than 3.
5. Speaks, understands and prints in English.
6. Gives written informed consent.

Exclusion Criteria for Detoxification Treatment Phase (DP)

1. Subjects mandated to treatment based upon a legal decision or as a condition of employment.
2. Subjects with evidence of substance dependence other than alcohol or nicotine dependence.
3. Subjects with psychosis or dementia at the time of the initial evaluation.
4. Female Subjects who are pregnant or lactating, or female Subjects of child bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include: tubal ligation, barrier (diaphragm or condom) with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection, and oral contraceptives.
5. Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator. EKG first degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <5 x ULN are acceptable), Subjects with impaired renal function as indicated by corrected creatinine clearance below 80 ml/min/70 kg as determined by the modified Cockcroft equation (CDC, 1986).
6. Subjects who have a positive urine drug screening (cocaine, amphetamines, opiates, barbiturates, benzodiazepines)
7. Subjects who have any disease of the gastrointestinal tract, liver or kidneys that could result in a possibility of altered metabolism or excretion of the study drug. As it is not possible to enumerate the many conditions which might impair absorption, metabolism, or excretion, the investigators will be guided by evidence such as: History of major gastrointestinal tract surgery (gastrectomy, gastrostomy, bowel resection, etc.) or a history of an active peptic ulcer or chronic disease of the GI tract, (ulcerative colitis, regional enteritis, or gastrointestinal bleeding).
8. Current unstable heart disease.
9. Known hypersensitivity to acamprosate.
10. Subjects taking psychotropic drugs (e.g., antidepressants, anxiolytic, antipsychotic, naltrexone, disulfiram, modafinil, stimulants and anticonvulsants) with the exception of oxazepam
11. Subjects receiving formal psychotherapy
12. Subjects having participated in any investigational drug trial within 30 days prior to the study.
13. Subjects with AIDS or other serious illnesses that may require hospitalization during the study.

Inclusion Criteria for Post-Detoxification Rehabilitative Treatment Phase (RP/Phase 2) with Open-Label Acamprosate

1. Has taken at least 5 days of acamprosate or placebo directly prior to initiating open-label acamprosate.
2. Successfully completed, within a 14-day period, outpatient detoxification. Successful completion of detoxification is defined as having a score of 1 or lower on the Clinical Institutes Withdrawal Assessment for Alcohol (CIWA; Shaw et al., 1981), and has at least 3 consecutive days of abstinence.
3. Has reduced medication taken specifically for detoxification (if applicable), i.e., oxazepam to 45 mg within 24-hour period prior to the post-detoxification rehabilitative treatment phase.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
1) the mean number of adverse events rated moderate to severe; | Phase I: up to 2 weeks
2) the week of detoxification treatment discontinuation; | Phase I: up to 2 weeks
3) the total amount of oxazepam given; | Phase I: up to 2 weeks
4) the rate of change in CIWA scores. | Phase I: up to 2 weeks
1) the mean number of adverse events rated moderate to severe; | Phase II: 10 weeks
2) the week of open-label treatment discontinuation; | Phase II: 10 weeks
3) any reemergence of detoxification symptoms; | Phase II: 10 weeks
4) % pills taken over what was proposed to be prescribed (medication exposure); | Phase II: 10 weeks
5) % days abstinent; | Phase II: 10 weeks
6) % days heavy drinking. | Phase II: 10 weeks

SECONDARY OUTCOMES:
Changes in alcohol craving will be measured by Penn Alcohol Craving Scale (PACS; Flannery et al, 1999) | 12 weeks
Changes in anxiety symptoms will be measured by the Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A; Hamilton, 1969) | 12 weeks
Changes in depressive symptoms will be measured by the Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D; Hamilton 1967) | 12 weeks
Changes in social functioning will be measured by several of the subscales of the Addiction Severity Index (ASI; McLellan et al, 1992); namely, medical, legal, psychiatric, and family/social. | 12 weeks
Quality of Life, measured by the Short Form-36 Health Status Questionnaire (SF-36; Ware & Sherbourne, 1999) | 12 weeks
Overall clinical impression of improvement will be measured by the Clinical Global Impression Scale (CGI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pettinati, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kampman KM, Pettinati HM, Lynch KG, Xie H, Dackis C, Oslin DW, Sparkman T, Sharkoski T, O'Brien CP. Initiating acamprosate within-detoxification versus post-detoxification in the treatment of alcohol dependence. Addict Behav. 2009 Jun-Jul;34(6-7):581-6. doi: 10.1016/j.addbeh.2009.03.014. Epub 2009 Mar 24. PMID 19345510